CLINICAL TRIAL: NCT05996003
Title: A Phase 2 Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of NS-089/NCNP-02 in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: NS-089/NCNP-02-201 in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NS-089/NCNP-02-201
Record Dates: First submitted 2023-07-18; First posted 2023-08-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy; Exon 44; DMD
Keywords: Exon 44 Skipping; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NS-089/NCNP-02 (Experimental): Experimental: NS-089/NCNP-02
  NS-089/NCNP-02 solution for infusion (Cohort 1)
  NS-089/NCNP-02 solution for infusion (Cohort 2)
  Interventions: Drug: NS-089/NCNP-02

INTERVENTIONS:
Drug: NS-089/NCNP-02 — Cohort 1:
  Part 1 Dose Level 1-3: a 4-week Treatment Phase at each treatment dose level
  Part 2 Single Dose Level: a 24-week Treatment Phase at the MTD of Part 1
  Cohort 2:
  Part 2 Single Dose Level: a 24-week Treatment Phase at the MTD of Part 1
  Other Names: Brogidirsen

SUMMARY:
This is a Phase 2, open-label, multi-center, 2-part study of NS-089/NCNP-02 administered by weekly IV infusion to ambulant boys aged ≥4 to <15 years with DMD due to mutations amenable to exon 44 skipping. Participants will receive a selected dose of NS-089/NCNP-02 administered once weekly.

The study consists of 2 parts: Part 1 and Part 2. Six participants (Cohort 1) will participate in both Part 1 and Part 2, and 14 participants (Cohort 2) will be added for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 4 years and <15 years of age
* Confirmed DMD mutation(s) in the dystrophin gene that is amenable to skipping of exon 44 to restore the dystrophin mRNA reading frame
* Able to walk independently without assistive devices
* Ability to complete the TTSTAND without assistance in <20 seconds
* Stable dose of glucocorticoid for at least 3 months and the dose is expected to remain on a stable dose for the duration of the study.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Has a body weight of <20 kg at the time of informed consent (applies to participants screening for Part 1 only)
* Evidence of symptomatic cardiomyopathy
* Current or previous treatment with anabolic steroids (e.g., oxandrolone) or products containing resveratrol or adenosine triphosphate within 3 months prior to first dose of study drug
* Current or previous treatment with any other investigational drug within 3 months prior to the first dose of study drug or within 5 times the half-life of a medication, whichever is longer
* Surgery within the 3 months prior to the first dose of study drug or planned during the study duration
* Previously treated in an interventional study of NS-089/NCNP-02
* Having taken any gene therapy.
* Having received exon skipping oligonucleotide within 1 year prior to the first dose of IP or is expected to receive exon skipping oligonucleotide prior to completion of study.
* Other exclusion criteria may apply.

Ages: 4 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Event and Adverse Drug Reaction | through study completion, up to follow-up phone call for Part 2
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Maximum plasma concentration (Cmax) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Time of the maximum plasma concentration (Tmax) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Terminal half-life (T1/2) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Area under the concentration-time curve from time 0 to the last time point (AUC0-t) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Area under the concentration-time curve from time 0 to infinity (AUC0-∞) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | [Time Frame: Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Total body clearance (CLtot) of NS-089/NCNP-02
Plasma pharmacokinetic (PK) parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] The volume in the terminal state (Vz) of NS-089/NCNP-02
Urine pharmacokinetic parameters | Day1, Week4 for each dose for Part 1, Day1 and Week24 for Part 2] Urinary excretion of NS-089/NCNP-02
Change from baseline in skeletal muscle dystrophin protein by immunoblot (Western blot). | Baseline, Week25

SECONDARY OUTCOMES:
Change from baseline in skeletal muscle dystrophin protein by mass spectrometry. | Baseline, Week25
Change from baseline in skeletal muscle dystrophin protein levels by immunofluorescence staining. | Baseline, Week25
Change from baseline in percentage of exon 44-skipped mRNA of skeletal muscle dystrophin | Baseline, Week25
North Star Ambulatory Assessment (NSAA) score | Baseline, Week13, Week25
  The NSAA is a functional scale devised for use in ambulant children with Duchenne muscular dystrophy (DMD). It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). It assesses abilities necessary to remain ambulant that have been found to progressively deteriorate in untreated DMD patients, as well as in other muscular dystrophies such as Becker Muscular Dystrophy. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
Time to Run/Walk 10 Meters (TTRW) | Baseline, Week13, Week25
Time to Stand (TTSTAND) | Baseline, Week13, Week25
Total distance of 6 Minute Walk Test (6MWT) | Baseline, Week13, Week25
Time to Climb 4 Stairs (TTCLIMB) | Baseline, Week13, Week25
Muscle strength measured by Quantitative Muscle Testing (QMT) | Baseline, Week13, Week25
Grip and pinch strength | Baseline, Week13, Week25
Performance of Upper Limb (PUL) 2.0. score | Baseline, Week13, Week25
  The PUL 2.0 provides both a total score and sub-scores for the 3 domains (shoulder, middle, and distal) that in DMD are progressively involved with a proximal to distal gradient. The PUL includes 22 items with an entry item to define the starting functional level. The 22 items are subdivided into the high-level shoulder dimension (6 items), middle level elbow dimension (9 items), and distal wrist and hand dimension (7 items). For weaker patients, a low score on the entry item (0-2) means high level items do not need to be performed. Scoring options vary across the scale between 0-1 and 0-2 according to performance. Each dimension can be scored separately with a maximum score of 12 for the high-level shoulder dimension, 17 for the middle level elbow dimension, and 13 for the distal wrist and hand dimension. A total score can be achieved by adding the 3 level scores (maximum total score of 42).

CONTACTS AND LOCATIONS:
Locations (22):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC - FL, Kissimmee, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - UT Southwestern/Children's Health, Dallas, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
- Japan (5):
  - Fukui Prefectural Hospital, Fukui-shi, Fukui
  - National Hospital Organization Nagara Medical Center, Nagara, Gifu-shi, Gifu
  - NHO Osaka Toneyama Medical Center, Toyonaka, Osaka
  - Shiga General Hospital, Moriyama-shi, Shiga
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
- Starship Children's Hospital, Auckland, New Zealand
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam
  - Seoul National University Hospital, Seoul
- Yeditepe University Kosuyolu Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Please follow this link for additional information on how to participate — https://mytomorrows.com/trials/discover-ns-089/en-us?utm_source=website&utm_medium=affiliate&utm_campaign=161_usa_en_web_organic_cnv_afi_link-for-ct-gov&utm_content=161_link-for-ct-gov_txt_link-for-ct-gov